CLINICAL TRIAL: NCT02338427
Title: Capacity of Amylose Characterisation Compare by Immunohistochemistry and Proteomic Analysis. Multicenter Prospective
Brief Title: Capacity of Amylose Characterisation Compare by Immunohistochemistry and Proteomic Analysis
Acronym: IPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHD 063-14
Record Dates: First submitted 2015-01-12; First posted 2015-01-14 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- proteomic (Experimental)
  Interventions: Other: Immunohistochemistry; Other: Proteomic analysis

INTERVENTIONS:
Other: Immunohistochemistry
Other: Proteomic analysis

SUMMARY:
Amyloidosis is involved in many rare diseases in relation to the diversity of amyloid proteins involved in the formation of abnormal tissue deposits. There are approximately 30 proteins involved in amylose's constitution. The therapeutic management varies depending on the type of amyloidosis observed.

The application of conventional techniques immunolabeling of amylose does not allow the comprehensive characterization of amylose forms, due to failures of the technic, the false positivity of some results, or lack of frozen tissue available for typing light chain (lambda, kappa).

In this study, the main objective is the comparison of two capacity of amylose characterisation: immunohistochemistry and proteomics analysis.

The purpose of this study is to validate the superiority of proteomic analysis by demonstrating the improvement of the precision, the reduction of technical failure, as well as the correction of erroneous diagnosis, authorizing a more adapted therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Upper age to 18 years
* Amylose diagnosis establish by tissue sample, after "Rouge Congo" coloration
* All patient with amylose identified by the two laboratory of anatomopathology
* Sample necessary for realized proteomic analysis
* No opposition at the participation of the study
* Patient sign an informed consent for biology collection

Exclusion Criteria:

* Tissue sample inadequate for apply immunohistochemistry or proteomic identification
* Patient trust, guardianship, under legal protection measure, deprived of freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-05; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Identification success of amylose by immunohistochemistry and proteomic analysis | Inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Hervé MAISONNEUVE, PH, Study Director — Centre Hospitalier Départementel Vendée
Locations (2):
- France (2):
  - Centre Hospitalier Departemental Vendee, La Roche-sur-Yon
  - CHU de Nantes, Nantes